CLINICAL TRIAL: NCT02195310
Title: The Use of PrevenaTM Incision Management System on Clean Closed Sternal Midline Incisions in Subjects at High Risk for Surgical Site Occurrences.
Brief Title: The Use of PrevenaTM on Clean Closed Sternal Midline Incisions in Subjects at High Risk for Surgical Site Occurrences.
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: due to futility
Sponsor: Solventum US LLC (Industry)
Collaborators: KCI Europe Holding B.V. (Industry); 3M (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KCI.2013.Prevena.01
Record Dates: First submitted 2014-07-16; First posted 2014-07-21 (Estimated); Results first posted 2019-08-05 (Actual); Last update posted 2024-10-02 (Actual); Status verified 2024-09

CONDITIONS: Surgical Site Occurences After Sternotomy; Wound Infection
Keywords: Sternotomy; Surgical site Occurences; Negative Pressure Wound Therapy; Surgical Site Infection
MeSH Terms: conditions — Wound Infection; Surgical Wound Infection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Prevena™ Incision Management System (Experimental): Subjects will receive sternal wound treatment in the operating room using Prevena™ Incision Management System according to the intended use
  Interventions: Device: Prevena™ Incision Management System
- Conventional sterile wound dressings (Active Comparator): Subjects will receive standard conventional wound therapy (SCWT) placed in the operating room, defined as using conventional sterile wound dressings (gauze).
  Interventions: Device: Conventional sterile wound dressings

INTERVENTIONS:
Device: Prevena™ Incision Management System — Prevena™ Incision Management System is used after sternotomy on the closed incision
  Other Names: Prevena Peel & Place
  Arms: Prevena™ Incision Management System
Device: Conventional sterile wound dressings — Conventional sterile wound dressings are placed after sternotomy on the closed incision
  Arms: Conventional sterile wound dressings

SUMMARY:
The purpose of this study is to compare the use of Prevena™ Incision Management System (IMS) versus standard wound care for the incision in subjects undergoing a sternal midline incision (sternotomy). The subjects targetted for the study are at high risk for surgical complications (like infections) around the environment of the incision.

The study is conducted in The Netherlands, Germany and Austria.

DETAILED DESCRIPTION:
The Prevena™ IMS is intended to manage the environment of closed surgically incision and surrounding intact skin for patients with an increased risk for developing post-operative complications such as infection.The purpose of this study is to compare the use of Prevena™ Incision Management System (IMS) versus standard wound care for the incision in subjects undergoing a sternal midline incision (sternotomy). The subjects targetted for the study are at high risk for surgical complications (like infections) around the environment of the incision.

The Prevena™ IMS is a small portable device, which consists of a mild vacuum unit that delivers negative pressure and a dressing that is intended for use over closed incisions after surgery. It is used for a minimum of 4 days up to a maximum of 7 days. This system is commercially available and has a CE mark, which means that it is approved for the use on the European market. It is intended to be applied immediately post sternotomy surgery on a closed clean incision.

The results of this study could contribute to a better and faster healing of the incision.

The study is conducted in The Netherlands, Germany and Austria.

ELIGIBILITY:
Inclusion Criteria:

* Is male or female and 18 years of age or older
* Is scheduled for elective cardiac surgery for which a median sternotomy is needed (including coronary artery bypass grafting (CABG), valvular repair or replacement with or without CABG). Elective surgery is defined as planned surgery a minimum of 24 hours before the procedure.
* Is capable of providing informed consent, which must be obtained prior to any study-related procedures
* Is willing and able to adhere to the study visit schedule and other protocol requirements.

Exclusion Criteria:

* Is pregnant
* The use of Prevena post surgery is contra indicated per investigator's discretion
* Has a systemic infection at the time of surgery: systemic infection is diagnosed on the basis of clinical signs of sepsis with or without a positive culture of an organism from the bloodstream
* Has a remote body site infection at the time of surgery (including dental, urinary or skin soft tissue infections)
* Is known to have a current nasal swab positive for methicillin-resistant staphylococcus aureus (MRSA)
* Has a known allergy or hypersensitivity to silver, or drape materials that contain acrylic adhesives
* Has a requirement for competing wound therapy and procedures.
* Any concomitant therapies (including other NPWT treatment) or procedures deviating from the clinical standard incision treatment or with investigational device at the location of the sternotomy (e.g. use of NPWT at other location of the body is allowed)
* Any other therapies or procedures that, in the opinion of the treating physician, would affect or influence postoperative wound stability or healing
* Is simultaneously participating in another interventional trial
* Requires use of liquid skin adhesives or glues during skin closure
* Is known to be serology positive for hepatitis B, hepatitis C or HIV

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 342 (Actual)
Dates: Start 2013-11-12 (Actual); Primary Completion 2016-08-15 (Actual); Study Completion 2016-10-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thanasie Markou, MD, PhD, Principal Investigator — Isala
Locations (13):
- Austria (3):
  - Medizinische Universitat Graz, Graz
  - Clinical Research Center Salzburg GmbH, Salzburg
  - Medizinische Universitaet Wien, Universitätsklinik für Chirurgie, Vienna
- Germany (5):
  - Deutsches Herzzentrum Berlin, Berlin
  - Charité Berlin, Berlin
  - Universitätsklinikum Erlangen, Erlangen
  - Westfälische Wilhelms-Universität Münster, Münster
  - Klinikum Nürnberg, Nuremberg
- Netherlands (5):
  - Catharina Ziekenhuis Eindhoven, Eindhoven, North Brabant
  - Isala Klinieken, Zwolle, Overijssel
  - Thoraxcentrum Research BV, Erasmus University Medical Center Rotterdam, Rotterdam, South Holland
  - Stichting St. Antonius ziekenhuis, Nieuwegein, Utrecht
  - University Medical Center Groningen, Groningen

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Prevena™ Incision Management System | Conventional Sterile Wound Dressings
Started | 173 | 169
Completed | 153 | 153
Not Completed | 20 | 16

BASELINE CHARACTERISTICS:
Groups:
- Prevena™ Incision Management System: Subjects will receive sternal wound treatment in the operating room with Prevena™ IMS according to the intended use
  Prevena™ Incision Management System: Prevena™ Incision Management System is used after sternotomy on the closed incision
- Total: Total of all reporting groups
Arm/Group | Prevena™ Incision Management System | Conventional Sterile Wound Dressings | Total
Number analyzed (Participants) | 173 | 169 | 342
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.1 (9.279) | 65.45 (10.304) | 66.29 (9.819)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 79 | 70 | 149
  Male | 94 | 99 | 193
Region of Enrollment [Number; unit: participants]
  Netherlands | 75 | 70 | 145
  Austria | 24 | 25 | 49
  Germany | 74 | 74 | 148

OUTCOME MEASURES:

1. Primary Outcome: Surgical Site Infection (SSI) Rate Within 34 Days Postoperatively, Defined as Superficial, Deep, and Organ/Space Infections as Per CDC Guidelines.
Description: The SSI rate (in %) was calculated for each treatment arm as follows:
  SSI rate = [Number of Subjects who experienced SSI] / [Number of Subjects Analyzed] * 100 Subjects included in the numerator for the SSI rate computation must have experienced an SSI post-surgery up to Day 30 (± 4 days). If a subject has the same SSI event on multiple occasions or experiences several events of other SSIs, the subject will be counted only once in the numerator for the first event
Time Frame: 30 ± 4 days
Population: Full Analysis Set: Included Subjects in the ITT Analysis Set that had no important disqualifying protocol deviations, who met the inclusion/exclusion criteria, and had completed SSI evaluations at visit 5 (Follow-up Day 30). Subjects were analyzed in the arm to which they were treated.
Measure: Number; unit: percentage of participants
Arm/Group | Prevena™ Incision Management System | Conventional Sterile Wound Dressings
Number analyzed (Participants) | 145 | 154
percentage of participants | 9.0 | 10.4
Statistical Analysis 1: Comparison: Prevena™ Incision Management System vs Conventional Sterile Wound Dressings; Test type: Superiority; p = 0.7007, Fisher Exact Test (2-sided)

ADVERSE EVENTS:
Arm/Group | Prevena™ Incision Management System | Conventional Sterile Wound Dressings
Serious Adverse Events (participants affected / at risk) | 63/173 | 55/169
Other Adverse Events (participants affected / at risk) | 85/173 | 96/169
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Prevena™ Incision Management System (N=173) | Conventional Sterile Wound Dressings (N=169)
Cardiac Tamponade (Cardiac disorders) | 8 | 3
Cardiogenic Shock (Cardiac disorders) | 4 | 2
Atrioventricular Block (Cardiac disorders) | 1 | 5
Pericardial Effusion (Cardiac disorders) | 3 | 1
Cardiac Failure (Cardiac disorders) | 0 | 4
Ventricular Failure (Cardiac disorders) | 2 | 1
Ventricular Fibrillation (Cardiac disorders) | 2 | 1
Ventricular Tachycardia (Cardiac disorders) | 2 | 1
Atrial Fibrillation (Cardiac disorders) | 1 | 1
Cardiac Arrest (Cardiac disorders) | 1 | 1
Cardiac Failure Congestive (Cardiac disorders) | 1 | 1
Right Ventricular Failure (Cardiac disorders) | 1 | 1
Myocardial Infarction (Cardiac disorders) | 0 | 2
Bundle Branch Block Left (Cardiac disorders) | 1 | 0
Cardiac Valve Disease (Cardiac disorders) | 1 | 0
Left Ventricular Failure (Cardiac disorders) | 1 | 0
Low Cardiac Output Syndrome (Cardiac disorders) | 1 | 0
Sick Sinus Syndrome (Cardiac disorders) | 1 | 0
Ventricular Flutter (Cardiac disorders) | 1 | 0
Angina Pectoris (Cardiac disorders) | 0 | 1
Bradycardia (Cardiac disorders) | 0 | 1
Electromechanical Dissociation (Cardiac disorders) | 0 | 1
Postoperative Infection (Infections and infestations) | 8 | 10
Pneumonia (Infections and infestations) | 3 | 3
Septic Shock (Infections and infestations) | 2 | 1
Groin Infection (Infections and infestations) | 2 | 0
Mediastinitis (Infections and infestations) | 1 | 1
Catheter Site Infection (Infections and infestations) | 0 | 2
Infection (Infections and infestations) | 0 | 2
Acute Endocarditis (Infections and infestations) | 1 | 0
Cystitis (Infections and infestations) | 1 | 0
Empyema (Infections and infestations) | 1 | 0
Pneumonia Bacterial (Infections and infestations) | 1 | 0
Respiratory Tract Infection (Infections and infestations) | 1 | 0
Abscess (Infections and infestations) | 0 | 1
Cellulitis (Infections and infestations) | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 1
Mediastinal Abscess (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 0 | 1
Wound Dehiscence (Injury, poisoning and procedural complications) | 6 | 9
Post Procedural Haemorrhage (Injury, poisoning and procedural complications) | 1 | 2
Dislocation of Sternum (Injury, poisoning and procedural complications) | 2 | 0
Haemothorax (Injury, poisoning and procedural complications) | 1 | 0
Rib Fracture (Injury, poisoning and procedural complications) | 1 | 0
Vascular Procedure Complication (Injury, poisoning and procedural complications) | 1 | 0
Wound Complication (Injury, poisoning and procedural complications) | 1 | 0
Wound Secretion (Injury, poisoning and procedural complications) | 1 | 0
Iatrogenic Injury (Injury, poisoning and procedural complications) | 0 | 1
Postoperative Thoracic Procedure Complication (Injury, poisoning and procedural complications) | 0 | 1
Spinal Fracture (Injury, poisoning and procedural complications) | 0 | 1
Haemodynamic Instability (Vascular disorders) | 4 | 2
Haematoma (Vascular disorders) | 2 | 1
Arterial Occlusive Disease (Vascular disorders) | 1 | 1
Haemorrhage (Vascular disorders) | 1 | 0
Ischaemia (Vascular disorders) | 1 | 0
Hypertensive Crisis (Vascular disorders) | 0 | 1
Vascular Insufficiency (Vascular disorders) | 0 | 1
Multi-Organ Failure (General disorders) | 2 | 2
Impaired Healing (General disorders) | 2 | 0
Chest Pain (General disorders) | 1 | 1
Sudden Cardiac Death (General disorders) | 1 | 0
Sudden Death (General disorders) | 0 | 1
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 4 | 2
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Apnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary Oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Cerebrovascular Accident (Nervous system disorders) | 4 | 1
Cerebral Infarction (Nervous system disorders) | 0 | 1
Dizziness (Nervous system disorders) | 0 | 1
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 1 | 0
Intestinal Haemorrhage (Gastrointestinal disorders) | 1 | 0
Large Intestine Perforation (Gastrointestinal disorders) | 1 | 0
Melaena (Gastrointestinal disorders) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Hypercreatininaemia (Metabolism and nutrition disorders) | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0
Malnutrition (Metabolism and nutrition disorders) | 0 | 1
Renal Insufficiency (Renal and urinary disorders) | 1 | 3
Delirium (Psychiatric disorders) | 2 | 1
Rehabilitation Therapy (Surgical and medical procedures) | 0 | 1
Removal of Foreign Body (Surgical and medical procedures) | 0 | 1
Leukocytosis (Blood and lymphatic system disorders) | 1 | 0
Amaurosis Fugax (Eye disorders) | 1 | 0
Anaphylactic Reaction (Immune system disorders) | 1 | 0
C-Reactive Protein Increased (Investigations) | 1 | 0
Prostatitis (Reproductive system and breast disorders) | 1 | 0
Skin Necrosis (Skin and subcutaneous tissue disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Prevena™ Incision Management System (N=173) | Conventional Sterile Wound Dressings (N=169)
Atrial Fibrillation (Cardiac disorders) | 45 | 43
Pericardial Effusion (Cardiac disorders) | 28 | 30
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 35 | 41
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 29 | 33
Wound Dehiscence (Injury, poisoning and procedural complications) | 24 | 19
Post Procedural Haematoma (Injury, poisoning and procedural complications) | 9 | 9
Postoperative Infection (Infections and infestations) | 7 | 9
Lung Infection (Infections and infestations) | 9 | 6
Oedema Peripheral (General disorders) | 7 | 12
Oedema (General disorders) | 9 | 5
Psychotic Disorder (Psychiatric disorders) | 12 | 14
Delirium (Psychiatric disorders) | 8 | 10
Diarrhoea (Gastrointestinal disorders) | 11 | 8
C-Reactive Protein Increased (Investigations) | 9 | 19
Anaemia (Blood and lymphatic system disorders) | 10 | 24
Wound Drainage (Surgical and medical procedures) | 10 | 5

LIMITATIONS AND CAVEATS:
Inclusion criteria were broad, expected event rates in the control group proved to be incorrect. Acelity plans to continue studying those at high risk for postoperative wound complications (e.g BMI>35).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes